CLINICAL TRIAL: NCT02358174
Title: Hemorrhoids and Metalloproteinases, Observational Study
Acronym: HeMe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Prof. Raffaele Serra, University of Catanzaro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ER.ALL.2013.27.A
Record Dates: First submitted 2015-01-22; First posted 2015-02-06 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: HEMORRHOIDS; Extracellular Matrix Alteration
Keywords: Hemorrhoids; MMP; NGAL; Matrix Metalloproteinases
MeSH Terms: conditions — Hemorrhoids | interventions — Hemorrhoidectomy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Experimental): Patients with symptomatic hemorrhoids - Grade I to IV sec. Goligher. Grade III to IV underwent Hemorrhoidectomy. Blood sampling for MMPs and NGAL plasma levels evaluation will be performed. Tissue sampling (obtained during hemorrhoidectomy) for MMPs and NGAL tissue levels evaluation will be performed in grade III-IV patients.
  Interventions: Procedure: Hemorrhoidectomy; Other: blood sampling; Other: tissue sampling
- Group II (Experimental): Healthy subjects without hemorrhoids as control groups for MMPs and NGAL plasma evaluation will be performed by means of Blood sampling.
  Interventions: Other: blood sampling

INTERVENTIONS:
Procedure: Hemorrhoidectomy — Grade III and IV patients were treated with surgery according to Milligan-Morgan (Milligan-Morgan laser optical fibers variant) procedure.
  All patients will perform blood sampling for MMPs and NGAL plasma levels evaluation
  Arms: Group I
Other: blood sampling — blood sampling for MMPs and NGAL plasma levels evaluation (ELISA test)
Other: tissue sampling — tissue sampling for MMPs and NGAL tissue levels evaluation (Western Blot)
  Arms: Group I

SUMMARY:
An association between hemorrhoidal disease and matrix metalloproteinases (MMPs) has been described previously. MMPs regulate extracellular structural proteins and tissue remodeling. Neutrophil gelatinase-associated lipocalin (NGAL) is involved in the regulation of MMP activity. The aim of this work was to study the relationship between the levels of MMPs and NGAL and different stages hemorrhoids.

The study provides potentially important insights to the understanding of the natural history of Hemorrhoids and MMPs and NGAL regulation.

DETAILED DESCRIPTION:
Introduction. An association between hemorrhoidal disease and matrix metalloproteinases (MMPs) has been described previously. MMPs regulate extracellular structural proteins and tissue remodeling. Neutrophil gelatinase-associated lipocalin (NGAL) is involved in the regulation of MMP activity. The aim of this work was to study the relationship between the levels of MMPs and NGAL and different stages hemorrhoids.

Methods. In a multicenter, open-label, prospective study, patients with hemorrhoids were recruited and represented the Group I (patients with symptomatic hemorrhoids - Grade I to IV sec. Goligher), a further group of healthy volunteer subjects were also recruited as the control group (Group II).

Enzyme-linked immunosorbent assay and Western blot analysis will evaluate the levels of immunoreactive MMPs and NGAL in all patients with hemorrhoids.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemorrhoids of both sex

Exclusion Criteria:

* Patients with cancer
* Hepatic failure
* Infectious or autoimmune diseases
* Arthritis
* Arterial aneurysms
* Hernias
* Chronic venous disease
* Nephritis, vascular ulcers, fibrosis, and other diseases associated with increased levels of MMPs were excluded from the study.
* Patients treated with corticosteroids or cytostatic drugs were also excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
MMPs and NGAL plasma and tissue levels measurement in patients with hemorrhoids | 15 months
  A new insight in the understanding of the natural history of. MMPs and NGAL play a role in development of disease and may represent molecular markers for the prevention of hemorrhoidal thrombosis.
  Unit of Measure: MMPs and NGAL plasma levels will be expressed as ng/mL. Tissue expression of MMPs and NGAL will be expressed as Arbitrary Units

REFERENCES:
- [Derived] Serra R, Gallelli L, Grande R, Amato B, De Caridi G, Sammarco G, Ferrari F, Butrico L, Gallo G, Rizzuto A, de Franciscis S, Sacco R. Hemorrhoids and matrix metalloproteinases: A multicenter study on the predictive role of biomarkers. Surgery. 2016 Feb;159(2):487-94. doi: 10.1016/j.surg.2015.07.003. Epub 2015 Aug 8. PMID 26263832